CLINICAL TRIAL: NCT04869111
Title: The BrainHealth Project, a Longitudinal Study in Generally Healthy Adults
Brief Title: The BrainHealth Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: University of Iowa (Other); University of California, Santa Barbara (Other); University of Kansas Medical Center (Other); Northeastern University (Other); Georgia State University (Other); University of Southern California (Other); Inova Health Care Services (Other); Methodist Healthcare (Other)
Responsible Party: Principal Investigator, Sandra Chapman, PhD, Professor, The University of Texas at Dallas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-745
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online SMART Intervention & Stress Solutions (Experimental): Strategic Memory Advanced Reasoning Training (SMART) teaches meta-cognitive strategies for individuals to apply to their daily lives for improved performance
  Interventions: Behavioral: Brain Health Training

INTERVENTIONS:
Behavioral: Brain Health Training — 1. On-line SMART - (Strategic Memory Advanced Reasoning Training) is a curriculum that teaches strategies of how to use the brain better, in such a way that may improve brain health and performance. SMART strives to achieve optimal cognitive function realized by the brain's ability to efficiently manage complex information by abstracting its essential meaning rather than attempting to memorize details, and to prioritize the information in order to attend to the most relevant parts.
  2. Stress Solutions - provides individuals with practical tools to enhance performance, reduce stress, build resilience and improve quality of life.
  3. Brain-Healthy Habits - daily reminders of habits you can track
  4. BrainHQ - participants will gain temporary access to the exercise-based cognitive training of BrainHQ after completing their 3rd BrainHealth Index

SUMMARY:
For an overview of the study and link TO REGISTER please go to -- https://brainhealth.utdallas.edu/programs/the-brainhealth-project/

The BrainHealth Project is a ten-year, longitudinal study focused on identifying determinants of brain health and performance. Participants will have the opportunity to complete semi-annual (twice a year) online assessments to track their performance over time. In between semi-annual assessments, participants will have access to online trainings and ongoing supplemental content regarding ways to optimize brain health and performance. Online one-on-one coaching sessions will be offered to participants to answer questions and provide support in applying the information to their daily lives. A small portion of participants will be invited to participate in the brain imaging portion of this study.

The main objectives are: (i) to characterize lifestyle, cognitive, and behavioral markers related to an individual's cognitive function from adolescent to elderly ages, (ii) to assess the neural/biological determinants predictive of maintenance of brain health, and (iii) to evaluate the impact of available cognitive and lifestyle interventions on improving and maintaining brain health and performance.

DETAILED DESCRIPTION:
Description of Study: For individuals who qualify to participate, they will be asked to complete online assessments and questionnaires twice a year. In between those time points, participants will participate in online trainings, exercises, and education regarding ways to optimize brain health, as well as overall health.

The assessments and trainings included in this protocol consist of the following:

Assessments:

BrainHealth Index (~90 min) - An online battery of cognitive measures and questionnaires. The Clarity section looks at complex thinking capacities such as reasoning, flexibility and strategy. In this section, you will be asked to complete different cognitive tasks. The questionnaires measure other aspects of life that relate to brain health, such as emotional well-being, quality of life, happiness, social support systems, and sleep. In this section, you will rate these aspects of your own life. Participants will also complete a 5 minute assessment with BrainHQ to measure processing speed.

The small group of participants who are invited to complete the brain imaging portion of the study will undergo annual brain imaging and will also complete brain gauge (in-person computer assessment). We will offer participants additional sub-studies, and they will have the opportunity to participate or not.

Online Trainings, habits, and resources:

Trainings can be accessed through the online dashboard and include videos, exercises, and application opportunities. Trainings include strategies to efficiently manage complex information by abstracting its essential meaning rather than attempting to memorize Training will also include strategies for stress management and healthy sleep routines, as well as other brain health education and resources. Most trainings are no more than 10 minutes a day.

Online Coaching:

Online coaching sessions will be offered to participants. Participants can elect to take advantage of this offer to the extent they chose.

For an overview of the study and LINK TO REGISTER please go to -- https://brainhealth.utdallas.edu/programs/the-brainhealth-project/

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Access to an internet connect and device
* Able to read information and hear sounds

Exclusion Criteria:

* Diagnosed neurodegenerative disease
* History of stroke, concussion, or brain injury that currently hinders you from functioning at your prior level
* Diagnosed with Autism Spectrum Disorder and not functioning independently

For an overview of the study and LINK TO REGISTER please go to -- https://brainhealth.utdallas.edu/programs/the-brainhealth-project/

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2038-08-01 (Estimated); Study Completion 2038-08-01 (Estimated)

PRIMARY OUTCOMES:
BrainHealth Index Score | Every 6 months for 10 years
  We will assess change on a holistic measure of cognitive, social, well-being, and daily life health on the BrainHealth Index (BHI) across multiple timepoints. Higher score = Better outcome)
Functional Magnetic Resonance Imaging (fMRI) Measure of Neural Correlations | Every 6 months for 10 years
  We will assess change in regional cerebral brain blood flow (using fMRI) in correlation with gains in complex abstraction across multiple timepoints. (higher correlation = better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra B Chapman, PhD, Principal Investigator — Center for BrainHealth
Locations (1):
- The Center for BrainHealth at The University of Texas at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chapman SB, Aslan S, Spence JS, Hart JJ Jr, Bartz EK, Didehbani N, Keebler MW, Gardner CM, Strain JF, DeFina LF, Lu H. Neural mechanisms of brain plasticity with complex cognitive training in healthy seniors. Cereb Cortex. 2015 Feb;25(2):396-405. doi: 10.1093/cercor/bht234. Epub 2013 Aug 28. PMID 23985135
- [Background] Chapman SB, Fratantoni JM, Robertson IH, D'Esposito M, Ling GSF, Zientz J, Vernon S, Venza E, Cook LG, Tate A, Spence JS. A Novel BrainHealth Index Prototype Improved by Telehealth-Delivered Training During COVID-19. Front Public Health. 2021 Mar 16;9:641754. doi: 10.3389/fpubh.2021.641754. eCollection 2021. PMID 33796498
- [Background] Chapman SB, Mudar RA. Enhancement of cognitive and neural functions through complex reasoning training: evidence from normal and clinical populations. Front Syst Neurosci. 2014 Apr 28;8:69. doi: 10.3389/fnsys.2014.00069. eCollection 2014. PMID 24808834
- [Background] Chapman SB, Aslan S, Spence JS, Keebler MW, DeFina LF, Didehbani N, Perez AM, Lu H, D'Esposito M. Distinct Brain and Behavioral Benefits from Cognitive vs. Physical Training: A Randomized Trial in Aging Adults. Front Hum Neurosci. 2016 Jul 18;10:338. doi: 10.3389/fnhum.2016.00338. eCollection 2016. PMID 27462210
- [Background] Chapman SB, Spence JS, Aslan S, Keebler MW. Enhancing Innovation and Underlying Neural Mechanisms Via Cognitive Training in Healthy Older Adults. Front Aging Neurosci. 2017 Oct 9;9:314. doi: 10.3389/fnagi.2017.00314. eCollection 2017. PMID 29062276
- [Background] Motes MA, Yezhuvath US, Aslan S, Spence JS, Rypma B, Chapman SB. Higher-order cognitive training effects on processing speed-related neural activity: a randomized trial. Neurobiol Aging. 2018 Feb;62:72-81. doi: 10.1016/j.neurobiolaging.2017.10.003. Epub 2017 Oct 12. PMID 29121545
- [Background] Han K, Davis RA, Chapman SB, Krawczyk DC. Strategy-based reasoning training modulates cortical thickness and resting-state functional connectivity in adults with chronic traumatic brain injury. Brain Behav. 2017 Apr 10;7(5):e00687. doi: 10.1002/brb3.687. eCollection 2017 May. PMID 28523229
- [Background] Vas A, Chapman S, Aslan S, Spence J, Keebler M, Rodriguez-Larrain G, Rodgers B, Jantz T, Martinez D, Rakic J, Krawczyk D. Reasoning training in veteran and civilian traumatic brain injury with persistent mild impairment. Neuropsychol Rehabil. 2016 Aug;26(4):502-31. doi: 10.1080/09602011.2015.1044013. Epub 2015 May 27. PMID 26018041
- [Background] Das N, Spence JS, Aslan S, Vanneste S, Mudar R, Rackley A, Quiceno M, Chapman SB. Cognitive Training and Transcranial Direct Current Stimulation in Mild Cognitive Impairment: A Randomized Pilot Trial. Front Neurosci. 2019 Apr 12;13:307. doi: 10.3389/fnins.2019.00307. eCollection 2019. PMID 31031581
- [Background] Han K, Martinez D, Chapman SB, Krawczyk DC. Neural correlates of reduced depressive symptoms following cognitive training for chronic traumatic brain injury. Hum Brain Mapp. 2018 Jul;39(7):2955-2971. doi: 10.1002/hbm.24052. Epub 2018 Mar 23. PMID 29573026
- [Background] Venza EE, Chapman SB, Aslan S, Zientz JE, Tyler DL, Spence JS. Enhancing Executive Function and Neural Health in Bipolar Disorder through Reasoning Training. Front Psychol. 2016 Nov 1;7:1676. doi: 10.3389/fpsyg.2016.01676. eCollection 2016. PMID 27847486
- [Background] Gallen CL, Baniqued PL, Chapman SB, Aslan S, Keebler M, Didehbani N, D'Esposito M. Modular Brain Network Organization Predicts Response to Cognitive Training in Older Adults. PLoS One. 2016 Dec 22;11(12):e0169015. doi: 10.1371/journal.pone.0169015. eCollection 2016. PMID 28006029